CLINICAL TRIAL: NCT01056796
Title: Compression Anastomosis For Low Anterior Resection in Previously Radiated Patients Using the CAR™ 27
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Niti Medical Technologies Ltd. (Industry)
Collaborators: University Hospital, Gasthuisberg (Other)
Responsible Party: Prof. Andre D'Hoore, Gasthuisberg University Hospital, Leuven, Belgium
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Version: January 6, 2010
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2010-01

CONDITIONS: Colorectal Cancer
Keywords: compression anastomosis; Colorectal cancer; Low anterior resection; Radiated to the pelvic area; Radiotherapy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CAR™ 27 (Experimental): Any patient with a diagnosis of colorectal cancer that has been previously radiated to the pelvic area (6-8 weeks prior to surgery) and that is electively scheduled for an open or laparoscopic total mesorectal excision (TME) and low anterior resection surgery (< 10cm from the anal verge) which requires the creation of an anastomosis, will be offered participation in this study.
  Interventions: Device: CAR™ 27

INTERVENTIONS:
Device: CAR™ 27 — Creation of a low colorectal (side or pouch low rectal) compression anastomosis in previously radiated patients
  Other Names: Compression Anastomosis Ring

SUMMARY:
The purpose of this study is:

Evaluation of the safety and effectiveness of the Compression Anastomosis Ring (CAR™ 27) device for creation of circular, colorectal anastomoses in previously radiated patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years old.
* Patient is scheduled for a non-emergency TME and low anterior resection (< 10cm from the anal verge).
* Patient has been radiated to the pelvic area 6-8 weeks prior to the study.
* Subject signs and dates a written informed consent form (ICF) and indicates an understanding of the study procedures.

Exclusion Criteria:

* Patient has known allergy to nickel.
* Patient undergoing an emergency procedure or has a diagnosis of bowel obstruction, bowel strangulation, peritonitis, bowel perforation, local or systemic infection, ischemic bowel, carcinomatosis or inflammatory bowel disease.
* Patients are participating in another clinical trial which may affect this study's outcomes.
* Patient has been taking regular steroid medication.
* Patient has contraindications to general anesthesia.
* Patient has preexisting sphincter problems or evidence of extensive local disease in the pelvis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
To evaluate for the occurrence of adverse events related to the use of the CAR™ 27 device, include anastomotic leak, bleeding, ring evacuation and strictures at 6 months. | Approx. 1 year

SECONDARY OUTCOMES:
Evaluation of the creation of a functioning CAR™ 27 anastomosis in radiated patients | Approx. 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Andre D'Hoore, Professor, Principal Investigator — Gasthuisberg University Hospital
Locations (1):
- University Hospital, Gasthuisberg, Leuven, Belgium